CLINICAL TRIAL: NCT03819738
Title: Functional Magnetic Resonance Imaging in Deep Brain Stimulation
Brief Title: fMRI in Deep Brain Stimulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S60058
Record Dates: First submitted 2019-01-22; First posted 2019-01-28 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy; Chronic Pain
Keywords: fMRI; epilepsy; pain; electrode; brain; neuromodulation; DBS
MeSH Terms: conditions — Epilepsy; Chronic Pain; Pain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: For each subject, condition effects will be estimated using the general linear model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fMRI intervention (Experimental)
  Interventions: Diagnostic Test: fMRI

INTERVENTIONS:
Diagnostic Test: fMRI — Functional MRI will be performed in 1 scan, which will take 1.5 h. (scanning time = 30 min)
  Other Names: DBS

SUMMARY:
With fMRI, we want to understand the mechanisms of brain neuromodulation in (dys)functional brain circuits, to obtain knowledge on involved brain networks in DBS.

DETAILED DESCRIPTION:
Deep brain stimulation represents a neurosurgical treatment option for specific refractory neurological and psychiatric disorders. In these patients a specific brain target is stimulated through an electrode with the use of an implantable pulse generator (IPG). In a functional MRI (fMRI) experiment, the investigators intend to perform imaging during stimulation ON and compare brain activations with the stimulation OFF condition. In this way, they aim to elucidate the involved brain network in deep brain stimulation. Since the connectivity of deep brain structures is complex, different activation patterns are expected in-between subjects and conditions. If specific activation patterns during the stimulation ON condition can be related to treatment response, this is of important clinical value. These findings can lead to an optimization of the deep brain target or even to different useful targets for brain stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Deep brain stimulation system implanted

Exclusion Criteria:

* Children and pregnant women will be excluded. Failure to follow to protocol is also an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-24 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Determine the functional networks that are involved in DBS | 5 years
  To determine differences in activations of functional networks between ON and OFF DBS in an fMRI experiment,
To link the involved network to outcome in DBS therapy | 5 years
  To link specific activation patterns during ON-OFF with a clinical value

CONTACTS AND LOCATIONS:
Overall Officials: Tom Theys, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Vlaams-Brabant, Belgium